CLINICAL TRIAL: NCT07175103
Title: Nurses' Self-Care Educational Programme (NSSCEP)
Brief Title: RCT to Evaluate the Efficacy of the NSSCEP in Reducing Burnout Among Jordanian Pediatric Oncology Nurses
Acronym: NSSCEP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Fadi Musa Yousef Abu Suqair, UNIVERSITI PUTRA MALAYSIA / Faculty of Medical and Health Science / Serdang, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 10/2025/10411; Prof Soh Kim Lam (Other: Universiti Putra Malaysia); Dr. Faiq Algbour (Other: Essra Hospital); IRB-JUH (Other: Jordan Unversity Hosptal); IRB (Other: Al Abdali Hospital)
Record Dates: First submitted 2025-08-26; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Paediatric Oncology; Nurses; Burnout; Occupational Stress; Self Care
MeSH Terms: conditions — Burnout, Psychological; Occupational Stress

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stress Self-Care Education Group (Experimental): Participants in this arm will receive the Nurses' Stress Self-Care Educational Program (NSSCEP), consisting of four educational sessions over one month focused on stress recognition, coping strategies, and resilience-building techniques. Participants will also complete weekly checklists and pre- and post-intervention surveys to assess burnout and stress levels.
  Interventions: Behavioral: Nurses' Stress Self-Care Educational Program (NSSCEP)
- Technical Skills Education Group (Placebo Comparator): Participants in this arm will receive a general technical skills program unrelated to stress management, delivered over one month in four sessions. Participants will also complete weekly checklists and pre- and post-intervention surveys to assess burnout and stress levels.
  Interventions: Other: General Technical Skills Program

INTERVENTIONS:
Behavioral: Nurses' Stress Self-Care Educational Program (NSSCEP) — A control intervention consisting of four 1-hour sessions over one month, focusing on general technical skills relevant to pediatric oncology nursing (e.g., procedural updates, equipment use). The program does not include stress management content. Participants complete weekly checklists and pre- and post-intervention surveys to measure burnout and stress levels.
  Arms: Stress Self-Care Education Group
Other: General Technical Skills Program — A control program with four 1-hour sessions over one month, focusing on technical skills (e.g., procedural updates, equipment use) without stress management content. Includes weekly checklists and pre/post surveys to measure burnout and stress.
  Arms: Technical Skills Education Group

SUMMARY:
The goal of this clinical trial is to learn if the Nurses' Stress Self-Care Educational Program (NSSCEP) can reduce burnout and occupational stress in Jordanian pediatric oncology nurses. The main questions it aims to answer are:

1. Does NSSCEP reduce symptoms of burnout in pediatric oncology nurses?
2. Does NSSCEP improve stress management skills among pediatric oncology nurses? Researchers will compare nurses participating in the NSSCEP to a control group receiving a general technical skills program to see if NSSCEP reduces burnout and improves stress management.

Participants will:

1. Attend four educational sessions over one month, focusing on stress recognition, coping strategies, and resilience-building techniques
2. Complete weekly checklists to track their application of stress management skills
3. Participate in pre- and post-intervention surveys to assess burnout and stress levels

DETAILED DESCRIPTION:
Burnout and occupational stress are significant challenges for pediatric oncology nurses in Jordan, who face intense emotional and professional demands while caring for critically ill children. The Nurses' Stress Self-Care Educational Program (NSSCEP) is designed to address this issue by equipping nurses with practical self-care strategies to enhance resilience and well-being. This study aims to evaluate the effectiveness of the NSSCEP in reducing burnout and stress levels among Jordanian pediatric oncology nurses working in hospital settings.

The NSSCEP is a structured, four-session educational intervention delivered over several weeks. Each session focuses on evidence-based self-care techniques, including stress management, mindfulness, emotional regulation, and coping strategies tailored to the unique challenges of pediatric oncology nursing. The program is facilitated by trained professionals and includes interactive workshops, group discussions, and practical exercises to foster skill development. The study compares the NSSCEP intervention group to a control group receiving standard workplace support to assess its impact on nurse well-being.

This trial addresses a critical gap in workplace interventions for Jordanian nurses, where cultural and systemic factors may influence stress and burnout. By implementing the NSSCEP, the study seeks to provide a scalable model for supporting nurse mental health in high-stress specialties. The findings may inform hospital policies and future interventions to promote sustainable nursing practice in Jordan and similar settings.

ELIGIBILITY:
Inclusion Criteria:

1. A registered nurse (RN) employed in a paediatric oncology unit in for at least 6 months.
2. Willingness to participate in all aspects of the study, including interventions, questionnaires, and follow-up assessments.
3. Ability to understand and communicate in English
4. Have ability Self-reported experience of burnout related to their role as a paediatric oncology nurse.
5. Nurses provide informed consent

Exclusion Criteria:

1. Less than six months of experience in paediatric oncology
2. Non-registered nurses (e.g., nursing assistants or technicians)
3. Non-voluntary participation or inability to provide informed consent
4. Inability to communicate in English
5. Involvement in leadership roles or administrative positions

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Reduction in Burnout Symptoms, improve Job satisfaction and missed nursing care | Pre-intervention (baseline) and post-intervention (at 4 weeks, following completion of the educational sessions).
  This study evaluates the Nurses' Stress Self-Care Educational Program (NSSCEP) for Jordanian pediatric oncology nurses. The four-week program includes workshops on stress management, mindfulness, and coping strategies to reduce burnout and enhance well-being. Burnout, job satisfaction, and missed nursing care are assessed using validated tools: Professional Quality of Life Scale, Nurse Job Satisfaction Scale, and MISSCARE Survey. Higher scores indicate better outcomes. The study aims to support nurse mental health and improve care quality in Jordanian hospitals.

CONTACTS AND LOCATIONS:
Overall Officials: Soh K Lam, Prof, Study Director — Universiti Putra Malaysia
Locations (1):
- Prince Hamza Hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wei H. The development of an evidence-informed Convergent Care Theory: Working together to achieve optimal health outcomes. Int J Nurs Sci. 2021 Dec 21;9(1):11-25. doi: 10.1016/j.ijnss.2021.12.009. eCollection 2022 Jan. PMID 35079601
- [Background] Wei H, Hardin SR, Watson J. A unitary caring science resilience-building model: Unifying the human caring theory and research-informed psychology and neuroscience evidence. Int J Nurs Sci. 2020 Nov 24;8(1):130-135. doi: 10.1016/j.ijnss.2020.11.003. eCollection 2021 Jan 10. PMID 33575453
- [Background] Wei H, Kifner H, Dawes ME, Wei TL, Boyd JM. Self-care Strategies to Combat Burnout Among Pediatric Critical Care Nurses and Physicians. Crit Care Nurse. 2020 Apr 1;40(2):44-53. doi: 10.4037/ccn2020621. PMID 32236429

DOCUMENTS (1):
  • Study Protocol (2025-08-22): https://cdn.clinicaltrials.gov/large-docs/03/NCT07175103/Prot_000.pdf